CLINICAL TRIAL: NCT06096909
Title: Early Initiation of Tafolecimab for Patients With Acute Coronary Syndromeundergoing Percutaneous Coronary Intervention in Chinese Population (EMPACT): A Randomized Controlled Trial
Brief Title: Early Initiation of Tafolecimab for Patients With Acute Coronary Syndromeundergoing Percutaneous Coronary Intervention in Chinese Population
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: China National Center for Cardiovascular Diseases (Other Government)
Collaborators: Innovent Biologics, Inc. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2021-CXGC03-002
Record Dates: First submitted 2023-09-28; First posted 2023-10-24 (Actual); Last update posted 2023-10-24 (Actual); Status verified 2023-10

CONDITIONS: Acute Coronary Syndrome; Non ST Segment Elevation Acute Coronary Syndrome
MeSH Terms: conditions — Acute Coronary Syndrome | interventions — Hydroxymethylglutaryl-CoA Reductase Inhibitors

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- experimental group (Experimental): intensive lipid lowering therapy
  Interventions: Drug: Tafolecimab; Drug: Statin
- control group (Active Comparator): conventional lipid lowering therapy
  Interventions: Drug: Cholesterol Absorption Inhibitor; Drug: Statin

INTERVENTIONS:
Drug: Tafolecimab — The PCSK9 mAb in this study is defined as Tafolecimab 150mg q2w subcutaneously. For the two groups of lipid-lowering regimens, the lipid-lowering drug regimens other than PCSK9 mAb were maintained throughout the study as much as possible in accordance with the guidelines related to blood lipids, provided that no serious safety problems occurred.
  Arms: experimental group
Drug: Cholesterol Absorption Inhibitor — Cholesterol absorption inhibitors (like Ezetimibe and Hybutimibe) are based on physician decisions, but need to be routinely dosed. Examples of Medications that Meet Study Requirements: Ezetimibe 10mg Po qd.
  Arms: control group
Drug: Statin — Statin are based on physician decisions, but need to be routinely dosed. Examples of Medications that Meet Study Requirements: Atorvastatin 20mg Po qn, Rosuvastatin 10mg Po qn or Pitavastatin 4mg Po qn.

SUMMARY:
For patients with ACS undergoing PCI, intensive lipid-lowering including PCSK9 monoclonal antibody should be started as soon as possible, that is, lower LDL-C level should be achieved as soon as possible. Compared with conventional lipid-lowering regimen, it is expected that the occurrence of major adverse cardiovascular events can still be reduced after drug discontinuation. Therefore, the optimization strategy of "for patients with ACS undergoing PCI, intensive lipid-lowering with PCSK9 monoclonal antibody can be started as soon as possible" is proposed.

DETAILED DESCRIPTION:
Atherosclerotic cardiovascular disease (ASCVD) is the leading cause of death worldwide, and its incidence is increasing yearly in China, which has not yet reached the inflection point. Acute coronary syndrome (ACS) is a severe form of ASCVD, and lipid-lowering and antithrombotic therapy are the two core therapies. In the latest ESC/EAS guidelines for lipid management, for ACS patients, the target LDL-C is <1.4 mmol/L and ≥50% reduction from baseline, and specific initiatives to achieve this target are proposed, emphasizing the timing of clinical application and status of the novel lipid-lowering agent-proprotein convertase subtilisin/kexin type 9 monoclonal antibody (PCSK9) (hereafter referred to as PCSK9 antibody). In recent years, large-scale randomized controlled trials and outcomes of PCSK9 antibodies have demonstrated that PCSK9 antibodies further reduce adverse cardiovascular events by significantly lowering LDL-C levels under the background statin (±cholesterol absorption inhibitor ) therapy. The introduction of PCSK9 antibodies allowed for the reduction of LDL-C to unprecedented levels. From the "cholesterol principle" perspective, it is theoretically reasonable to add a PCSK9 inhibitor to statins as soon as possible during hospitalization for ACS patients. Still, there is no clear evidence from large RCTs. Current evidence supports that for ACS patients, PCSK9 antibodies could be used only when LDL-C is still not up to standard based on treatment with the maximum tolerable dose of statins during the first 2-3 months. However, the immediate initiation of PCSK9 antibodies during the acute phase of ACS (before hospital discharge) has yet to be studied.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 to 75 years;
* clinical diagnosis with non-ST-segment elevation acute coronary syndrome (NSTE-ACS) ;
* undergoing PCI
* baseline LDL-C 1.8 mmol/L 3.4 mmol/L note: NSTE-ACS includes non-ST-elevation myocardial infarction and unstable angina.

Exclusion Criteria:

* Severe heart failure (Killip III or IV) or cardiogenic shock;
* Previous hemorrhagic cerebrovascular disease history;
* Uncontrolled or recurrent arrhythmic events;
* poorly controlled hypertension;
* Severe hepatic and renal insufficiency (ALT/AST> 3 times upper limit of normal, eGFR<30 ml/kg/1.73m2, or ongoing dialysis) or creatine kinase elevation>5 times upper limit of normal
* malignant tumor;
* Intolerance to statins or cholesterol absorption inhibitors;
* Intolerance to injections;
* Life expectancy <1 year;
* poor compliance.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3684 (Estimated)
Dates: Start 2023-11-01 (Estimated); Primary Completion 2025-11-01 (Estimated); Study Completion 2027-11-01 (Estimated)

PRIMARY OUTCOMES:
Major adverse cardiovascular and cerebrovascular events (MACCE) | at the end of 2 years
  Including cardiovascular death, non-fatal myocardial infarction, non-fatal stroke, hospitalization for unstable angina, and coronary revascularization). The coronary revascularization includes coronary intervention (PCI), coronary artery bypass grafting (CABG).

SECONDARY OUTCOMES:
major adverse cardiovascular events (MACEs) | at the end of 6 months
  Cardiovascular death, nonfatal myocardial infarction, hospitalization for unstable angina, and coronary revascularization.
Major adverse cardiovascular and cerebrovascular events (MACCE) | at the end of 1 years
  Including cardiovascular death, non-fatal myocardial infarction, non-fatal stroke, hospitalization for unstable angina, and coronary revascularization). The coronary revascularization includes coronary intervention (PCI), coronary artery bypass grafting (CABG).

OTHER OUTCOMES:
Additional observed endpoint 1 | at the end of 2 years
  Cardiovascular death
Additional observed endpoint 2 | at the end of 2 years
  non-fatal myocardial infarction
Additional observed endpoint 3 | at the end of 2 years
  non-fatal stroke
Additional observed endpoint 4 | at the end of 2 years
  hospitalization for unstable angina
Additional observed endpoint 5 | at the end of 2 years
  coronary revascularization

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-08-25): https://cdn.clinicaltrials.gov/large-docs/09/NCT06096909/Prot_SAP_000.pdf
  • Informed Consent Form (2023-08-25): https://cdn.clinicaltrials.gov/large-docs/09/NCT06096909/ICF_001.pdf